CLINICAL TRIAL: NCT03042104
Title: Evaluation of Transcatheter Aortic Valve Replacement Compared to Surveillance for Patients With Asymptomatic Severe Aortic Stenosis
Brief Title: EARLY TAVR: Evaluation of TAVR Compared to Surveillance for Patients With Asymptomatic Severe Aortic Stenosis
Acronym: EARLY TAVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-07
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Heart Diseases; Aortic Stenosis, Severe
Keywords: Aortic valve; Asymptomatic; Transcatheter aortic valve replacement
MeSH Terms: conditions — Heart Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TAVR (Experimental): Transcatheter aortic valve replacement (TAVR)
  Interventions: Device: Edwards SAPIEN 3 / SAPIEN 3 Ultra THV
- CS (No Intervention): Clinical surveillance (CS)

INTERVENTIONS:
Device: Edwards SAPIEN 3 / SAPIEN 3 Ultra THV — Patients will receive the SAPIEN 3 / SAPIEN 3 Ultra THV.
  Other Names: SAPIEN 3, SAPIEN 3 Ultra
  Arms: TAVR

SUMMARY:
This study will evaluate the safety and effectiveness of the Edwards SAPIEN 3/SAPIEN 3 Ultra Transcatheter Heart Valve (THV) compared with clinical surveillance (CS) in asymptomatic patients with severe, calcific aortic stenosis.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multicenter study. Patients will be randomized to receive either transcatheter aortic valve replacement (TAVR) with the Edwards SAPIEN 3 / SAPIEN 3 Ultra THV or clinical surveillance. Patients will be stratified by whether they are able to perform a treadmill stress test. Patients who have a positive stress test will be followed in a registry to collect data on subsequent treatment and mortality, as applicable.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. Severe aortic stenosis
3. Patient is asymptomatic
4. LV ejection fraction ≥ 50%
5. Society of Thoracic Surgeons (STS) risk score ≤ 10
6. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Patient is symptomatic
2. Patient has any concomitant valvular, aortic, coronary artery disease requiring surgery making AVR a Class I indication.
3. Native aortic annulus size unsuitable for sizes 20, 23, 26, or 29 mm THV
4. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
5. Left ventricular outflow tract calcification that would increase the risk of annular rupture or significant paravalvular leak post TAVR
6. Evidence of an acute myocardial infarction ≤ 30 days before randomization
7. Aortic valve is unicuspid, bicuspid with unfavorable features for TAVR, or is non-calcified
8. Severe aortic regurgitation (>3+)
9. Severe mitral regurgitation (>3+) or ≥ moderate mitral stenosis
10. Pre-existing mechanical or bioprosthetic valve in any position
11. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of randomization
12. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy, or hypercoagulable states
13. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of randomization
14. Hypertrophic cardiomyopathy with obstruction
15. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
16. Inability to tolerate or condition precluding treatment with anti-thrombotic therapy
17. Stroke or transient ischemic attack within 90 days of randomization
18. Renal insufficiency and/or renal replacement therapy
19. Active bacterial endocarditis within 180 days of randomization
20. Severe lung disease or currently on home oxygen
21. Severe pulmonary hypertension
22. History of cirrhosis or any active liver disease
23. Significant frailty as determined by the Heart Team
24. Significant abdominal or thoracic aortic disease that would preclude safe passage of the delivery system
25. Patient refuses blood products
26. BMI >50 kg/m2
27. Estimated life expectancy <24 months
28. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
29. Currently participating in an investigational drug or another device study.
30. Active SARS-CoV-2 infection (Coronavirus-19 [COVID-19]) or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 901 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
All-cause death, all stroke, and unplanned cardiovascular hospitalization | When all patients have reached 2-year follow-up
  The number of patients that have any of these conditions

SECONDARY OUTCOMES:
Composite of 1) alive, 2) Kansas City Cardiomyopathy Questionnaire (KCCQ) score ≥75 and 3) KCCQ decrease ≤10 points | 2 years
  The number of patients that meet all of these criteria
Left Ventricular Health | 2 years
  Echocardiographic measurements that will assess the health of the left ventricle
Change in Left Ventricular Ejection Fraction (LVEF) | 2 years
  The average change in LVEF from baseline
New onset atrial fibrillation | When all patients have reached 2-year follow-up
  The number of patients that develop this condition
Death or disabling stroke | When all patients have reached 2-year follow-up
  The number of patients that have any of these conditions

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Généreux, MD, Principal Investigator — Gagnon Cardiovascular Institute - Morristown Medical Center, Cardiovascular Research Foundation
Locations (77):
- United States (74):
  - Banner University Medical Center, Phoenix, Arizona
  - Mills Peninsula Health Services, Burlingame, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Huntington Hospital, Pasadena, California
  - UC Davis Medical Center, Sacramento, California
  - Kaiser San Francisco Medical Center, San Francisco, California
  - Stanford Hospital and Clinics Palo Alto, Stanford, California
  - UC Health Northern Colorado (Medical Center of the Rockies), Loveland, Colorado
  - Yale University, New Haven, Connecticut
  - Washington Hospital Center DC, Washington D.C., District of Columbia
  - The Cardiac & Vascular Institute Research Foundation, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center Chicago, Chicago, Illinois
  - NorthShore University HealthSystem Research Institution, Evanston, Illinois
  - Alexian Brothers Hospital Network, Lisle, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart, Saint Cloud, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Atlantic Health System Hospital Corp - Morristown Medical Center, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Rutgers Robert Wood Johnson Medical School, Piscataway, New Jersey
  - Albany Medical College, Albany, New York
  - University at Buffalo - Kaleida Health, Buffalo, New York
  - NYU Langone Hosptial - Long Island, Mineola, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - Cornell University, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolina's Health System, Charlotte, North Carolina
  - NC Heart and Vascular (Rex Hospital), Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel Health System, Columbus, Ohio
  - The Ohio Health Research Institute, Columbus, Ohio
  - Kaiser Portland, Clackamas, Oregon
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Allegheny - Singer Research Institute, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Heart Hospital Baylor Plano, Dallas, Texas
  - Texas Health Physician Group, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Intermountain Medical Center Salt Lake City, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart and Vascular Institute (Fairfax Inova), Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Providence Everett, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Hamilton Health Sciences, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genereux P, Schwartz A, Pibarot P, Lindman BR, Cohen DJ, Oldemeyer JB, Fearon WF, Babaliaros V, Daniels D, Chhatriwalla AK, Suradi HS, Shah PB, Szerlip M, Mack MJ, Dahle T, Goel K, O'Neill WW, Davidson CJ, Makkar RR, Sheth T, Williams M, Russo MJ, Guerrero M, McCabe J, Leipsic J, Zhao Y, Hahn RT, Blanke P, Leon MB. Outcomes of Early vs Delayed Aortic Valve Replacement: Analysis of the EARLY TAVR Valve Implant Population. JACC Cardiovasc Interv. 2025 Nov 24;18(22):2761-2773. doi: 10.1016/j.jcin.2025.09.029. PMID 41297989
- [Derived] Lindman BR, Pibarot P, Schwartz A, Cohen DJ, Giustino G, Oldemeyer JB, Strote JA, Babaliaros V, Devireddy CM, Fearon WF, Fischbein MP, Daniels D, Spies C, Chhatriwalla AK, Kavinsky CJ, Shah P, Szerlip M, Dahle T, Stegman B, O'Leary JM, O'Neill WW, Makkar RR, Davidson CJ, Sheth T, DeVries JT, Southard J, Depta JP, Pop A, Leipsic J, Blanke P, Li Y, Hahn RT, Leon MB, Genereux P. Left Ventricular Health and TAVR Timing in Asymptomatic Severe Aortic Stenosis: Analysis From the EARLY TAVR Trial. J Am Coll Cardiol. 2025 Sep 7:S0735-1097(25)07642-9. doi: 10.1016/j.jacc.2025.08.071. Online ahead of print. PMID 41128701
- [Derived] Lindman BR, Pibarot P, Schwartz A, Oldemeyer JB, Su YR, Goel K, Cohen DJ, Fearon WF, Babaliaros V, Daniels D, Chhatriwalla A, Suradi HS, Shah P, Szerlip M, Mack MJ, Dahle T, O'Neill WW, Davidson CJ, Makkar R, Sheth T, Depta J, DeVries JT, Southard J, Pop A, Sorajja P, Hahn RT, Zhao Y, Leon MB, Genereux P; EARLY TAVR Trial Executive Committee and Study Investigators. Cardiac Biomarkers in Patients With Asymptomatic Severe Aortic Stenosis: Analysis From the EARLY TAVR Trial. Circulation. 2025 Jun 3;151(22):1550-1564. doi: 10.1161/CIRCULATIONAHA.125.074425. Epub 2025 Mar 31. PMID 40163596
- [Derived] Genereux P, Schwartz A, Oldemeyer JB, Pibarot P, Cohen DJ, Blanke P, Lindman BR, Babaliaros V, Fearon WF, Daniels DV, Chhatriwalla AK, Kavinsky C, Gada H, Shah P, Szerlip M, Dahle T, Goel K, O'Neill W, Sheth T, Davidson CJ, Makkar RR, Prince H, Zhao Y, Hahn RT, Leipsic J, Redfors B, Pocock SJ, Mack M, Leon MB; EARLY TAVR Trial Investigators. Transcatheter Aortic-Valve Replacement for Asymptomatic Severe Aortic Stenosis. N Engl J Med. 2025 Jan 16;392(3):217-227. doi: 10.1056/NEJMoa2405880. Epub 2024 Oct 28. PMID 39466903
- [Derived] Genereux P, Schwartz A, Oldemeyer B, Cohen DJ, Redfors B, Prince H, Zhao Y, Lindman BR, Pibarot P, Leon MB. Design and rationale of the evaluation of transcatheter aortic valve replacement compared to surveillance for patients with asymptomatic severe aortic stenosis: The EARLY TAVR trial. Am Heart J. 2024 Feb;268:94-103. doi: 10.1016/j.ahj.2023.11.019. Epub 2023 Dec 4. PMID 38056546
- [Derived] Zelis JM, Tonino PAL, Pijls NHJ, De Bruyne B, Kirkeeide RL, Gould KL, Johnson NP. Coronary Microcirculation in Aortic Stenosis: Pathophysiology, Invasive Assessment, and Future Directions. J Interv Cardiol. 2020 Jul 22;2020:4603169. doi: 10.1155/2020/4603169. eCollection 2020. PMID 32774184